CLINICAL TRIAL: NCT03602976
Title: A Single-center, Open Label, Cross-over Study on the Effects of Ursodeoxycholic Acid (UDCA) in Patients With Hepatic Sarcoidosis
Brief Title: Ursodeoxycholic Acid (UDCA) for Hepatic Sarcoidosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to adequately recruit subjects in COVID-19 pandemic
Sponsor: Ethan Weinberg (Other)
Collaborators: American Association for the Study of Liver Diseases (Other); Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ethan Weinberg, Assistant Professor of Clinical Medicine, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 828780
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Hepatic Sarcoidosis, Elevated Alkaline Phosphatase
Keywords: hepatic sarcoidosis; elevated alp
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: Subjects will act as their own controls by undergoing a six-month initial observational period prior to initiating the six-month UDCA intervention
Masking Description: All subjects will receive appropriately dosed UDCA after six months of observation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Observation (No Intervention)
- UDCA at Month 6 (Experimental)
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — weight-based dosing
  Other Names: UDCA; ursodiol
  Arms: UDCA at Month 6

SUMMARY:
This study aims to (1) evaluate efficacy of UDCA in improving liver function and quality of life; (2) monitor safety, tolerability of UDCA, as well as progression of hepatic sarcoidosis and liver disease, in patients diagnosed with hepatic sarcoidosis. A minimum of 10 subjects will be followed for 12 months. For all subjects, initial 6 months will be observational; in subsequent 6 months, UDCA will be administered. Visits will occur every 3 months and involve routine blood collection.

DETAILED DESCRIPTION:
Sarcoidosis is a relatively rare, poorly defined autoimmune disease characterized by the formation of sterile granulomas in affected organs, including the liver. The diagnosis of hepatic sarcoid is often presumed based upon an elevated liver-specific isoenzyme of alkaline phosphatase or imaging findings suggestive of portal hypertension, hepatomegaly, or liver lesions in a patient with known pulmonary sarcoidosis; a minority of hepatic sarcoid cases are diagnosed through liver biopsy. The mainstay of treatment of systemic sarcoidosis in those with symptoms is immunosuppression with corticosteroids, which are gradually tapered over months. The disease course for sarcoidosis can vary; patients who are asymptomatic can be monitored without therapy, while some require intermittent corticosteroids for flares. The expert guidelines for treatment of hepatic sarcoid suggest waiting until a patient is symptomatic or experiencing evidence of liver dysfunction to treat. This approach is in opposition to the treatment of primary liver diseases in which treatment is often initiated based upon abnormal lab values even without symptoms, as symptoms of liver disease (ascites, variceal bleeding, pruritus, jaundice, and encephalopathy) often occur late in the disease. The approach to the treatment of hepatic sarcoid should be similar to two other autoimmune liver diseases: autoimmune hepatitis (AIH) and primary biliary cholangitis (PBC). Liver decompensation can be prevented in both AIH and PBC if the disease is diagnosed and treated in the early stages. The first-line treatment for AIH is immunosuppression with corticosteroids and azathioprine; for PBC, it is Ursodeoxycholic acid (UDCA). In a similar vein, patients with hepatic sarcoid may benefit from earlier initiation of therapy. Given its excellent safety profile and minimal side effects, UDCA may be the consensus first-line treatment for hepatic sarcoid, a disease that, like PBC, usually causes a cholestatic liver injury. There have been case reports and retrospective studies documenting the beneficial effects of UDCA on hepatic sarcoid. However, thus far, there have been no clinical trials to evaluate the efficacy of UDCA in hepatic sarcoid. This pilot study will examine the effects of UDCA in a small sample of patients at the University of Pennsylvania. Patients with a prior diagnosis of sarcoidosis and lab/imaging findings suggestive of hepatic sarcoid would be approached. The primary endpoint is a reduction in alkaline phosphatase from baseline. Secondary endpoints include safety and tolerability of UDCA, new or worsening symptoms of hepatic sarcoidosis and liver disease, changes in bilirubin and transaminases, and liver stiffness as measured by Fibroscan. A minimum of ten patients will be enrolled for a twelve-month study with the total study time of two years. It is hypothesized that UDCA will lead to modest decreases in alkaline phosphatase levels in patients with hepatic sarcoid with minimal side effects. Overtime a long-term decline in alkaline phosphatase could decrease the risk of hepatic decompensation in patients with hepatic sarcoid.

As an exploratory objective and optional sub-study, the investigators will include the methacetin breath test (MBT), a noninvasive tool to assess microsomal capacity to metabolize the nonradioactive compound 13-Carbon-labeled Methacetin. The MBT will be used in parallel with clinical and laboratory parameters (Fibroscan, liver enzymes) to assess subjects liver function prior to and following intervention with UDCA. Changes in the methacetin breath tests in all subjects prior to and following intervention with UDCA will be examined as a secondary exploratory endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Systemic sarcoidosis with evidence of liver involvement as denoted by any of the following:

   * Elevated liver-specific alkaline phosphatase
   * Granulomas on liver biopsy
   * Hepatomegaly on imaging
   * Portal Hypertension (via imaging or endoscopy)
2. Stable dose of immunosuppressant, if taking (no dose variation for 6 months)
3. If cirrhotic, absence of hepatocellular carcinoma as indicated by imaging within 6 months of screening

Exclusion Criteria:

1. Female who is pregnant, planning to become pregnant during the study, or breastfeeding
2. Clinically significant abnormalities, co-morbidities, or recent alcohol/drug abuse that make the subject an unsuitable candidate
3. Concurrent liver disease including hepatitis B, hepatitis C, alcohol-related liver disease, autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis
4. Currently on UDCA
5. Prior intolerance to UDCA
6. Receipt of any investigational product within a time period equal to 10 half-lives of the product, or 6 weeks (whichever is longer), to study drug administration
7. Current evidence of hepatic decompensation (variceal bleeding, hepatic encephalopathy, or ascites). In the event potential participant is post-transplant, no evidence of hepatic decompensation since transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UDCA at Month 6
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Number of subjects that completed observation period of 6 months
Groups:
- Subjects That Completed 6-month Observation Period: Single-Arm UDCA
Arm/Group | Subjects That Completed 6-month Observation Period
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 58 [50 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Alkaline Phosphatase (U/L) [Mean (Full Range); unit: U/L] | 257.7 [113 to 428]
Gamma Glutamyl Transferase (U/L) [Mean (Full Range); unit: U/L] | 302.5 [64 to 814]
Liver Stiffness by Transient Elastography [Mean (Full Range); unit: kPa] — (Fibroscan, kPa) Population: One baseline subject did not undergo fibroscan at baseline assessment due to COVID restrictions
  kPa
    number analyzed (Participants) | 5
    (all) | 8.3 [4.6 to 14.3]
Bilirubin [Mean (Full Range); unit: mg/dL] | 0.72 [0.4 to 1.2]
Alamine Aminotransferase (ALT) [Mean (Full Range); unit: U/L] | 50.8 [24 to 103]
Aspartate Aminotransferase (AST) [Mean (Full Range); unit: U/L] | 43.3 [21 to 66]

OUTCOME MEASURES:

1. Primary Outcome: Alkaline Phosphatase (U/L) or Gamma Glutamyl Transferase (U/L) 6 Months After Initiation of Ursodeoxycholic Acid
Description: Alkaline Phosphatase (U/L) or Gamma Glutamyl Transferase (U/L) 6 months after initiation of ursodeoxycholic acid
Time Frame: 6 months after initiaiton of UDCA
Measure: Mean (Full Range); unit: U/L
Arm/Group | UDCA at Month 6
Number analyzed (Participants) | 6
U/L
  Alkaline Phosphatase | 202.2 [128 to 321]
  Gamma Glutamyl Transferase | 111.8 [25 to 304]
Statistical Analysis 1: Comparison: UDCA at Month 6; For GGT; Test type: Superiority; p = 0.059, t-test, 2 sided; Mean Difference (Final Values) = 190.7
Statistical Analysis 2: Comparison: UDCA at Month 6; For Alkaline Phosphatase; Test type: Superiority; p = 0.23, t-test, 2 sided; Mean Difference (Final Values) = 55.5

2. Secondary Outcome: Liver Stiffness
Description: kPa as assessed by Fibroscan
Time Frame: Baseline and 6 months after initiation of UDCA
Measure: Mean (Full Range); unit: kPa
Groups:
- Observation: Completed observation and had fibroscan at time of completion
Arm/Group | Observation | UDCA at Month 6
Number analyzed (Participants) | 5 | 5
kPa | 8.3 [4.6 to 14.3] | 6.3 [3.7 to 13.2]
Statistical Analysis 1: Comparison: UDCA at Month 6; Test type: Superiority; p = 0.36, t-test, 2 sided; Mean Difference (Final Values) = 2.06

3. Secondary Outcome: Bilirubin
Time Frame: Baseline and 6 months after initiation of UDCA
Measure: Mean (Full Range); unit: mg/dL
Groups:
- Observation: Completed observation
Arm/Group | Observation | UDCA at Month 6
Number analyzed (Participants) | 6 | 6
mg/dL | 0.72 [0.4 to 1.2] | 0.77 [0.3 to 1.9]
Statistical Analysis 1: Comparison: UDCA at Month 6; Test type: Superiority; p = 0.73, t-test, 2 sided; Mean Difference (Final Values) = 0.05

4. Secondary Outcome: AST
Time Frame: Baseline and 6 months after initiation of UDCA
Measure: Mean (Full Range); unit: U/L
Arm/Group | Observation | UDCA at Month 6
Number analyzed (Participants) | 6 | 6
U/L | 43.3 [21 to 66] | 31.2 [18 to 47]
Statistical Analysis 1: Comparison: UDCA at Month 6; Test type: Superiority; p = 0.094, t-test, 2 sided; Mean Difference (Final Values) = 12.2

5. Secondary Outcome: ALT
Time Frame: Baseline and 6 months after initiation of UDCA
Measure: Mean (Full Range); unit: U/L
Arm/Group | Observation | UDCA at Month 6
Number analyzed (Participants) | 6 | 6
U/L | 50.8 [24 to 103] | 29.8 [15 to 62]
Statistical Analysis 1: Comparison: UDCA at Month 6; Test type: Superiority; p = 0.11, t-test, 2 sided; Mean Difference (Final Values) = 21

ADVERSE EVENTS:
Time Frame: Entirety of the study - up to 2 years
Arm/Group | UDCA at Month 6
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UDCA at Month 6 (N=7)
Nausea (Gastrointestinal disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination due to poor recruitment in light of the COVID-19 pandemic, affecting data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT03602976/Prot_SAP_000.pdf